CLINICAL TRIAL: NCT01526135
Title: Multicentric Randomized Phase III Trial Comparing Adjuvant Chemotherapy With Gemcitabine Versus 5-fluorouracil, Leucovorin, Irinotecan and Oxaliplatin (mFolfirinox) in Patients With Resected Pancreatic Adenocarcinoma
Brief Title: Trial Comparing Adjuvant Chemotherapy With Gemcitabine Versus mFolfirinox to Treat Resected Pancreatic Adenocarcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: Canadian Cancer Trials Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Prodige 24 / Accord 24; NCIC CTG PA.6 (Other: NCIC); 2011-002026-52 (EudraCT Number)
Record Dates: First submitted 2012-02-01; First posted 2012-02-03 (Estimated); Last update posted 2022-01-04 (Actual); Status verified 2022-01

CONDITIONS: Pancreatic Adenocarcinoma (Ductal Adenocarcinoma)
Keywords: National multicentric phase III superiority trial
MeSH Terms: interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A GEMCITABINE (Active Comparator): Arm A : Gemcitabine 1000 mg/m² IV infusion over 30 minutes, weekly, during 3 weeks + 1 week of rest (= 1 cycle) repeated 6 times (i.e., 6 cycles) during 24 weeks
  Interventions: Drug: Gemcitabine
- Arm B mFOLFIRINOX (Experimental): Arm B : mFOLFIRINOX every 14 days, 12 cycles, 24 weeks. Oxaliplatin (Eloxatin®) 85 mg/m² D1 over 2 hours, followed by Irinotecan (Campto®) 150 mg/m² D1 over 90 minutes to begin 30 min. after the Folinic acid infusion is started.
  Folinic acid 400 mg/m² (racemic mixture) (or 200 mg/m² if L-folinic acid is used), IV infusion over 2 hours.
  5-FU 2.4 g/m² IV continuous infusion over 46 hours (1200 mg/m²/ day)
  Interventions: Drug: mFolfirinox

INTERVENTIONS:
Drug: mFolfirinox — mFolfirinox every 14 days, 12 cycles, 24 weeks.
  mFolfirinox : Oxaliplatin (Eloxatin®) 85 mg/m² D1 over 2 hours, followed by Irinotecan (Campto®) 150 mg/m² D1 over 90 minutes to begin 30 min. after the Folinic acid infusion is started.
  Folinic acid 400 mg/m² (racemic mixture) (or 200 mg/m² if L-folinic acid is used), IV infusion over 2 hours.
  5-FU 2.4 g/m² IV continuous infusion over 46 hours (1200 mg/m²/ day)
  Arms: Arm B mFOLFIRINOX
Drug: Gemcitabine — Gemcitabine 1000 mg/m² IV infusion over 30 minutes, weekly, during 3 weeks + 1 week of rest (= 1 cycle) repeated 6 times (i.e., 6 cycles) during 24 weeks
  Arms: Arm A GEMCITABINE

SUMMARY:
This is a multicentric randomized phase III trial comparing adjuvant chemotherapy with gemcitabine versus 5-fluorouracil, leucovorin, irinotecan and oxaliplatin (mFolfirinox) in patients with resected pancreatic adenocarcinoma.

DETAILED DESCRIPTION:
STUDY DESIGN/ Evaluation criteria Main criterion: efficacy The main criterion is the disease-free survival at 3 years. Disease-free survival is the time delay between the date of randomization and the date at which the 1st cancer-related event such as local relapse, distant metastasis, a second cancer or death from any cause is observed. Patients without event at the time of anlaysis will be censored at the date of last follow-up visit.

Locoregional relapse is a disease relapse occurring at the site of primary resection, in the pancreas or in the associated regional lymph nodes.

Metastatic relapse is the distant disease recurrence involving any possible sites of relapse (peritoneal, hepatic, pulmonary, and distant lymph nodes).

Secondary criteria Overall and specific survival Overall survival is the time delay between the date of randomization and the patient's death, irrespective of its cause. Patients who are still living at the time of analysis will be censored at the date of last follow-up visit.

Specific survival is the time delay between the date of randomization and the patient's death due to the treated cancer or a treatment-related complication.

Metastasis-free survival Metastasis-free survival is the time delay between the date of randomization and the date of the 1st distant event occurrence (peritoneal, hepatic, pulmonary, and lymph nodes). Loco-regional events will be discarded and patients still living without metastasis at the time of analysis will be censored at the date of last follow-up examination objectively assessing this type of event.

Tolerance Patients evaluable for toxicity must have received at least one course or injection of the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven pancreatic ductal adenocarcinoma. Intraductal papillary mucinous tumor of the pancreas (IPMT) with invasive components are eligible.
2. Macroscopically complete resection (R0 or R1 resection).
3. Patients aged from 18 to 79 years.
4. WHO performance status 0-1.
5. No prior radiotherapy and no previous chemotherapy.
6. Full recovery from surgery and patient able to receive chemotherapy: adequate oral nutrition of ≥1500 calories per day and free of significant nausea and vomiting.
7. Adequate hematologic function (Absolute neutrophil count ANC ≥1,500 cells/mm³, platelets ≥100 000 cells/mm³ and hemoglobin ≥10 g/L - possibly after transfusion -).
8. Serum total bilirubin ≤1.5 times the institutional upper limit of normal.
9. Creatinine level <130 micromol/L (14.7 mg/L).
10. Patient of child-bearing potential (for female patient: study entry after a menstrual period and a negative pregnancy test) must agree to use two medically acceptable methods of contraception (one for the patient and one for the partner) during the study and for 4 months after the last study treatment intake for women and 6 months for men.
11. Interval since surgery between 21 and 84 days.
12. Patient information and signed informed consent.
13. Public or private health insurance coverage.

Exclusion Criteria:

1. Other types of non-ductal tumor of the pancreas, including endocrine tumors or acinar cell adenocarcinoma, cystadenocarcinoma and malignant ampulloma.
2. Metastases (including ascites or malignant pleural effusion).
3. Macroscopic incomplete tumor removal (R2 resection).
4. CA 19-9 > 180 U/ml within 21 days of registration on study.
5. No heart failure or coronary heart disease symptoms.
6. No major comorbidity that may preclude the delivery of treatment or active infection (HIV or chronic hepatitis B or C) or uncontrolled diabetes.
7. Pre-existing neuropathy, Gilbert's disease or genotype UGT1A1 * 28 / * 28.
8. Inflammatory disease of the colon or rectum, or occlusion or sub-occlusion of the intestine or severe postoperative uncontrolled diarrhea.
9. Concomitant occurrence of another cancer, or history of cancer except in situ carcinoma of the cervix treated or basal cell carcinoma or squamous cell carcinoma.
10. Fructose intolerance.
11. Persons deprived of liberty or under guardianship.
12. Psychological, familial, sociological or geographical condition potentially. hampering compliance with the study protocol and follow-up schedule.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 493 (Actual)
Dates: Start 2012-04-16 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2021-07-16 (Actual)

PRIMARY OUTCOMES:
disease-free survival (DFS) | 3 YEARS
  to compare disease-free survival (DFS) at 3 years between the experimental and control arms.

SECONDARY OUTCOMES:
Overall survival | 36 MONTHS
Specific survival | 36 MONTHS

CONTACTS AND LOCATIONS:
Overall Officials: Thierry CONROY, PROF, Principal Investigator — Centre Alexis Vautrin-VANDOEUVRE LES NANCY
Locations (52):
- Canada (19):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - CancerCare Manitoba, St. Boniface General Hospital, Winnipeg, Manitoba
  - Dr Leon Richard Oncology Centre, Moncton, New Brunswick
  - The Royal Victoria Hospital - Cancer Care Program, Barrie, Ontario
  - Department of Medical Oncology Health Sciences North, Greater Sudbury, Ontario
  - Juravinski Cancer centre at Hamilton Health Sciences, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston General Hospital, Kingston, Ontario
  - Ottawa Health Research Institute, Ottawa, Ontario
  - Niagara Health System, St. Catharines, Ontario
  - General Surgery - TGH Site, Univ. Health Network, Toronto, Ontario
  - CHUM - Hopital Notre-Dame, Montreal, Quebec
  - McGill University (Department of Oncology), Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec
  - Allain Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, University of Saskatchewan, Saskatoon, Saskatchewan
  - The Moncton Hospital, Moncton
  - CHUQ - Hotel-Dieu de Quebec, Québec
  - Algoma District Cancer Program, Sault Area Hospital, Sault Ste. Marie
- France (33):
  - CHU Nord, Amiens
  - ICO Paul Papin, Angers
  - Hôpital Avicenne, Bobigny
  - Institut Bergonié, Bordeaux
  - CHU Côte de Nacre, Caen
  - Hôpital Beaujon, Clichy
  - Hôpital Louis Pasteur, Colmar
  - CHU de Dijon - Site Bocage, Dijon
  - CHD Vendée, La Roche-sur-Yon
  - Hôpital Huriez, Lille
  - Centre Léon Bérard, Lyon
  - Hôpital de la Croix-Rousse, Lyon
  - Hôpital Privé Jean Mermoz, Lyon
  - CHU Nord, Marseille
  - CHU Timone Adulte, Marseille
  - Fondation Ambroise Paré / Hôpital Européen, Marseille
  - Institut Paoli Calmettes, Marseille
  - CH Layné, Mont-de-Marsan
  - CHU De ST Eloi, Montpellier
  - CRCL Val d'Aurelle, Montpellier
  - Centre Antoine-Lacassagne, Nice
  - CHR Orléans - La Source, Orléans
  - Groupe Hospitalier Paris Saint Joseph, Paris
  - Groupe Hospitalier Pitié-Salpêtrière, Paris
  - Hôpital Saint-Jean, Perpignan
  - Hôpital Haut-Lévêque, Pessac
  - Centre hospitalier de Reims, Reims
  - CHU Rouen, Rouen
  - Centre René Gauducheau, Saint-Herblain
  - Centre Paul Strauss, Strasbourg
  - Hôpital Trousseau, Tours
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Hôpital de Brabois-CHU de Nancy, Vandœuvre-lès-Nancy

REFERENCES:
- [Derived] Conroy T, Castan F, Lopez A, Turpin A, Ben Abdelghani M, Wei AC, Mitry E, Biagi JJ, Evesque L, Artru P, Lecomte T, Assenat E, Bauguion L, Ychou M, Bouche O, Monard L, Lambert A, Hammel P; Canadian Cancer Trials Group and the Unicancer-GI-PRODIGE Group. Five-Year Outcomes of FOLFIRINOX vs Gemcitabine as Adjuvant Therapy for Pancreatic Cancer: A Randomized Clinical Trial. JAMA Oncol. 2022 Nov 1;8(11):1571-1578. doi: 10.1001/jamaoncol.2022.3829. PMID 36048453
- [Derived] Conroy T, Hammel P, Hebbar M, Ben Abdelghani M, Wei AC, Raoul JL, Chone L, Francois E, Artru P, Biagi JJ, Lecomte T, Assenat E, Faroux R, Ychou M, Volet J, Sauvanet A, Breysacher G, Di Fiore F, Cripps C, Kavan P, Texereau P, Bouhier-Leporrier K, Khemissa-Akouz F, Legoux JL, Juzyna B, Gourgou S, O'Callaghan CJ, Jouffroy-Zeller C, Rat P, Malka D, Castan F, Bachet JB; Canadian Cancer Trials Group and the Unicancer-GI-PRODIGE Group. FOLFIRINOX or Gemcitabine as Adjuvant Therapy for Pancreatic Cancer. N Engl J Med. 2018 Dec 20;379(25):2395-2406. doi: 10.1056/NEJMoa1809775. PMID 30575490